CLINICAL TRIAL: NCT02048943
Title: A Phase Ib Study of Dovitinib in Combination With Gemcitabine and Nab-Paclitaxel in Patients With Advanced Solid Tumors and Pancreatic Cancer
Brief Title: Dovitinib Lactate, Gemcitabine Hydrochloride, and Paclitaxel Albumin-Stabilized Nanoparticle Formulation in Treating Patients With Advanced Solid Tumors or Pancreatic Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 242513; NCI-2014-00119 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 242513 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH)
Record Dates: First submitted 2014-01-27; First posted 2014-01-29 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Duct Cell Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage III Pancreatic Cancer; Stage IV Pancreatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one; Gemcitabine; Taxes; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (dovitinib, gemcitabine, nab-paclitaxel) (Experimental): Patients receive dovitinib lactate PO QD 5 days per week, paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: dovitinib lactate; Drug: gemcitabine hydrochloride; Drug: paclitaxel albumin-stabilized nanoparticle formulation; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: dovitinib lactate — Given PO
  Other Names: CHIR-258; receptor tyrosine kinase inhibitor TKI258; RTK inhibitor TKI258; TKI258
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Drug: paclitaxel albumin-stabilized nanoparticle formulation — Given IV
  Other Names: ABI-007; nab paclitaxel; nab-paclitaxel; nanoparticle albumin-bound paclitaxel
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the highest and safest doses of dovitinib lactate, paclitaxel albumin-stabilized nanoparticle formulation, and gemcitabine hydrochloride when given together. Dovitinib lactate disrupts the activity of fibroblast growth factor receptors and reduces cancer growth and spread. Gemcitabine hydrochloride and paclitaxel albumin-stabilized nanoparticle formulation are anti-cancer drugs for treating many cancer types.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose and recommended phase II dose of dovitinib (dovitinib lactate) when administered concurrently with gemcitabine (gemcitabine hydrochloride) and nab-paclitaxel (paclitaxel albumin-stabilized nanoparticle formulation) in patients with advanced solid malignancies.

II. To characterize the safety profile of dovitinib, gemcitabine and nab-paclitaxel combination in patients with advanced solid malignancies.

SECONDARY OBJECTIVES:

I. To characterize the pharmacokinetic profile of dovitinib, nab-paclitaxel, gemcitabine and their metabolites when administered concurrently in patients with advanced solid malignancies.

II. To determine the preliminary efficacy of the study combination in patients with advanced solid tumors and pancreas adenocarcinoma.

III. To explore serum and tumor biomarkers predictive of efficacy to the study combination.

OUTLINE: This is a dose-escalation study of dovitinib lactate.

Patients receive dovitinib lactate orally (PO) once daily (QD) 5 days per week, paclitaxel albumin-stabilized nanoparticle formulation intravenously (IV) over 30 minutes, and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Part A and Part B2: Histologically or cytologically confirmed solid tumors that are advanced or metastatic that gemcitabine and/or nab-paclitaxel containing treatment is considered a rational option
* Part Bl: Histologically or cytologically confirmed adenocarcinoma of the pancreas that is locally advanced or metastatic
* Part Bl: At least one malignant lesion not previously irradiated that can be safely biopsied, and patient is agreeable to undergo fresh tumor biopsy
* Patients with at least one measurable site of disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1 that has not been previously irradiated
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Life expectancy >= 3 months
* Absolute neutrophil count (ANC) >= 1,500 cells/mm^3 (SI units 1.5 x 10^9/L)
* Platelets >= 100,000 cells/mm^3 (SI units 100 x 10^9/L)
* Hemoglobin >= 9 g/dL (SI units 90 g/L)
* Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/serum glutamate pyruvate transaminase (SGPT) =< 1.5 x upper limit of normal (ULN)
* Bilirubin =< 1.5 x ULN
* Serum creatinine =< 1.5 x ULN
* International normalized ratio (INR) =< 1.5 (anticoagulation is allowed if target INR =< 1.5 on a stable dose of warfarin or on a stable dose of LMW heparin for > 2 weeks at the first dose of study agent)
* If urinalysis shows proteinuria, 24 hour urine collection is to be performed and the 24 hour urine protein is to be < 2 grams to be eligible
* Willing and able to comply with scheduled visits, treatment plan and laboratory tests
* Ability to understand and willingness to sign a written informed consent; a signed informed consent must be obtained prior to any study specific procedures

Exclusion Criteria:

* Patients who have received the last administration of an anti-cancer therapy including chemotherapy, immunotherapy, hormonal therapy and monoclonal antibodies (but excluding nitrosourea, mitomycin-C, targeted therapy and radiation) =< 4 weeks prior to starting study drug, or who have not recovered from side effects of such therapy
* Patients who have received the last administration of nitrosourea or mitomycin-C =< 6 weeks prior to starting study drug, or who have not recovered from the side effects of such therapy
* Patients who have received targeted therapy (e.g., sunitinib, sorafenib, pazopanib) =< 2 weeks prior to starting study drug, or who have not recovered from the side effects of such therapy
* Patients who have had radiotherapy =< 4 weeks prior to starting study drug, or =< 2 weeks prior to starting study drug in the case of localized radiotherapy (e.g., for analgesic purpose or for lytic lesions at risk of fracture), or who have not recovered from radiotherapy toxicities
* Patients who have undergone major surgery (e.g., intra-thoracic, intra-abdominal or intrapelvic), open biopsy or significant traumatic injury =< 4 weeks prior to starting study drug, or patients who have had minor procedures, percutaneous biopsies or placement of vascular access device =< 1 week prior to starting study drug, or who have not recovered from side effects of such procedure or injury
* Impaired cardiac function or clinically significant cardiac diseases, including any of the following:

  * History or presence of serious uncontrolled ventricular arrhythmias or presence of serious uncontrolled atrial fibrillation,
  * Clinically significant resting bradycardia
  * Known left ventricular ejection fraction (LVEF) assessed by 2-dimensional (2-D) echocardiogram (ECHO) < 50% or lower limit of normal (whichever is higher) or multiple gated acquisition scan (MUGA) < 45% or lower limit of normal (whichever is higher),
  * Any of the following within 6 months prior to study entry: myocardial infarction (MI), severe/unstable angina, coronary artery bypass graft (CABG), congestive heart failure (CHF), cerebrovascular accident (CVA), transient ischemic attack (TIA), pulmonary embolism (PE)
  * Uncontrolled hypertension defined by a systolic blood pressure (SBP) >= 160 mmHg and/or diastolic blood pressure (DBP) >= 100 mm Hg, with or without anti-hypertensive medication
* Previous pericarditis; clinically significant pleural effusion in the previous 12 months or current ascites requiring two or more interventions/month
* Any active gastrointestinal (GI) impairment which, in the opinion of the investigator, would impair or alter the absorption of dovitinib (e.g., ulcerative colitis, or Crohn's disease)
* Positive hemoccult test result within 14 days prior to the start of study treatment
* Cirrhosis, chronic active hepatitis or chronic persistent hepatitis
* Known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory)
* Patients who are currently receiving oral anticoagulation treatment with therapeutic doses of warfarin with goal INR > 1.5; patients receiving anticoagulation by subcutaneous injection such as heparin, enoxaparin, fondaparinux that are not expected to interact with study medications will be eligible
* History of alcoholism, drug addiction, or any psychiatric or psychological condition which, in the opinion of the investigator, would impair study compliance
* Uncontrolled diarrhea >= Common Terminology Criteria for Adverse Events (CTCAE) grade 2
* Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g., active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol
* Pregnant or breast-feeding women
* Women of child-bearing potential, defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (e.g., who has had menses any time in the preceding 12 consecutive months), must have a negative serum pregnancy test =< 3 days prior to starting study treatment
* Women of child-bearing potential, who are biologically able to conceive, not employing 2 forms of highly effective contraception; male not using at least at least one form of highly effective contraception will be excluded; highly effective contraception (e.g., male condom with spermicide, diaphragm with spermicide, intra-uterine device) must be used by both sexes during the study and must be continued for 8 weeks after the end of study treatment; oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study
* Patients with known brain metastases or who have signs/symptoms attributable to brain metastases and have not been assessed with radiologic imaging to rule out the presence of brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of dovitinib lactate, defined as the highest dose level at which < 33% of patients experience study treatment-related dose-limiting toxicity, graded using the National Cancer Institute (NCI) CTCAE version 4.0 | 28 days
Incidence of adverse events graded by NCI CTCAE version 4.0 | Up to 4 weeks
  Characterized by type, frequency, timing, seriousness and relationship to study treatment. All toxicities and adverse events will be summarized with frequencies and descriptive measures, and tabulated according to body system, severity and relation to treatment. Demographic data and baseline disease characteristics will be displayed, and summary statistics will be used to describe patient population.

SECONDARY OUTCOMES:
Plasma pharmacokinetic (PK) parameters of dovitinib lactate | Pre-dose, 0.5, 1-2,4-5, 6-8, 24 hours post-dose day 1 of course 2; pre-dose trough day 8 of course 2
  Pharmacokinetic parameters will be summarized for each cohort of patients. Comparison of PK parameters among the dose levels will be performed using non-parametric statistical methods for K-independent samples. Drug-drug interaction will be examined comparing PK parameters using nonparametric statistical methods.
Plasma PK parameters of gemcitabine hydrochloride | Prior to end of infusion, and 0.5, 1-2, and 4-6 hours post-end of infusion day 1 of course 2; prior to infusion of IV chemotherapy day 8 of course 2
  Pharmacokinetic parameters will be summarized for each cohort of patients. Comparison of PK parameters among the dose levels will be performed using non-parametric statistical methods for K-independent samples. Drug-drug interaction will be examined comparing PK parameters using nonparametric statistical methods.
Plasma PK parameters of paclitaxel albumin-stabilized nanoparticle formulation | Prior to end of infusion, and 0.5, 1-2, and 4-6 hours post-end of infusion day 1 of course 2; prior to infusion of IV chemotherapy day 8 of course 2
  Pharmacokinetic parameters will be summarized for each cohort of patients. Comparison of PK parameters among the dose levels will be performed using non-parametric statistical methods for K-independent samples. Drug-drug interaction will be examined comparing PK parameters using nonparametric statistical methods.
Survival (expansion cohort) | 6 months
  Overall survival will be estimated using Kaplan-Meier method.
Response rate, defined according to RECIST 1.1 (expansion cohort) | Up to 4 weeks
Progression-free survival (expansion cohort) | Up to 4 weeks
Biomarker expression levels in tumor specimens | Baseline
  Differences in biomarkers between responders and non-responders will be explored with frequencies and summary statistics. Tests for differences in continuously measured biomarkers will be done with standard two-sample testing procedures. Categorical biomarkers will be tested with Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Wee Ma, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States